CLINICAL TRIAL: NCT00369421
Title: Diagnosis and Treatment of Patients With Inborn Errors of Metabolism or Other Genetic Disorders
Brief Title: Diagnosis and Treatment of Patients With Inborn Errors of Metabolism
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 760238; 76-HG-0238
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-11-24

CONDITIONS: Arterial Calcification Due to Deficiency of CD73
Keywords: Biochemical Diseases; Rare Diseases; Family Studies; Screening; Next Generation Sequencing; Natural History
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Healthy Volunteers
- Patients: Patients with unique disorders
- Unaffected family members: Unaffected family members of patients

SUMMARY:
Researchers intend on diagnosing and treating certain inborn errors of metabolism. By doing this researchers hope to expand their knowledge about these disorders and provide access to patients of interest for research, teaching, and clinical experience.

Patients participating in this study will be examined and treated on an out patient basis, if practical. However, patients requiring specialized tests or treatments will be admitted to the NIH Clinical Center as necessary. Researchers will use only accepted medical procedures in diagnosing (medical history, physical examinations, X-ray studies, eye examinations, blood tests, and urine tests) and treating the patients involved in this study. Additional tests may be required on a case to case basis.

Many patients seen in this study will go on to be enrolled in a specific disease-related research study.<TAB>

DETAILED DESCRIPTION:
Study Description:

We propose to characterize the etiology and natural history of rare inborn errors of metabolism and other genetic disorders, both known and yet-to-be discovered. In so doing, we will expand our knowledge about these disorders and provide access to patients of interest for research, teaching, and clinical experience.

Objectives:

The overall aim of this protocol is to advance our knowledge of genetic disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants 1 month or older will have been or will be referred to this protocol with a known or suspected inborn error of metabolism, heritable disorder, or genetic predisposition. Participants over two years of age will be admitted only if they are medically stable and require admission to the Clinical Center for diagnosis. Children ages 1 month to 2 years or under 12 kg will be reviewed by the Pediatric Consult Service prior to scheduling and if approved will be evaluated.

Examples of disorders that will be under this protocol include inherited developmental defects or diatheses toward infections, cancer, or an environmentally induced disease. The principal investigator, along with consulting specialists, will review the medical records of prospective participants and offer admission based upon the potential to help the individual, to learn from the participant, or to initiate clinical or basic research suggested by the participant s workup. This protocol is not intended to serve as an umbrella protocol for small studies of specific disorders. In general, no more than 5 families known to have the same disorder will be investigated under this protocol.

Some participants will be relatives of patients with known diagnoses, and their specimens will be obtained for the purpose of heterozygote testing or to serve as controls to help diagnose the proband. All participants shall be seen as inpatients, outpatients or via Telehealth at the discretion of the principal investigator, based upon particular research interests and expertise. Normal adult volunteers aged 18 years or older will be enrolled to provide control blood and urine specimens.

EXCLUSION CRITERIA:

* Participants under 1 month of age will not be seen at the NIH Clinical center because care is more readily proffered to older individuals at the Clinical Center.
* Participants over two years of age will not be admitted if they are medically unstable and do not require admission to the Clinical Center for diagnosis.
* Pregnant women are excluded.

Ages: 1 Month to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Unique disorders.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 1978-09-12 (Actual)

PRIMARY OUTCOMES:
Clinical phenotyping | years to decades followup
  Clinical characterization.

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
pending
Supporting Information: Study Protocol
Time Frame: pending
Access Criteria: pending

REFERENCES:
- [Background] Gahl WA, Adamson M, Kaiser-Kupfer I, Ludwig IH, O'Connell HJ, Cohen W, Barranger J. Biochemical phenotyping of a single sibship with both cystinosis and Fabry disease. J Inherit Metab Dis. 1985;8(3):127-31. doi: 10.1007/BF01819297. PMID 3027448
- [Background] Bernardini I, Rizzo WB, Dalakas M, Bernar J, Gahl WA. Plasma and muscle free carnitine deficiency due to renal Fanconi syndrome. J Clin Invest. 1985 Apr;75(4):1124-30. doi: 10.1172/JCI111806. PMID 3988933
- [Background] Kaiser-Kupfer MI, Caruso RC, Minkler DS, Gahl WA. Long-term ocular manifestations in nephropathic cystinosis. Arch Ophthalmol. 1986 May;104(5):706-11. doi: 10.1001/archopht.1986.01050170096030. PMID 3518682
- [Derived] Theng EH, Brewer CC, Oheim R, Zalewski CK, King KA, Delsmann MM, Rolvien T, Gafni RI, Braddock DT, Jeffrey Kim H, Ferreira CR. Characterization of hearing-impairment in Generalized Arterial Calcification of Infancy (GACI). Orphanet J Rare Dis. 2022 Jul 19;17(1):273. doi: 10.1186/s13023-022-02410-w. PMID 35854274
- [Derived] Cohen JI, Manoli I, Dowdell K, Krogmann TA, Tamura D, Radecki P, Bu W, Turk SP, Liepshutz K, Hornung RL, Fassihi H, Sarkany RP, Bonnycastle LL, Chines PS, Swift AJ, Myers TG, Levoska MA, DiGiovanna JJ, Collins FS, Kraemer KH, Pittaluga S, Jaffe ES. Hydroa vacciniforme-like lymphoproliferative disorder: an EBV disease with a low risk of systemic illness in whites. Blood. 2019 Jun 27;133(26):2753-2764. doi: 10.1182/blood.2018893750. Epub 2019 May 7. PMID 31064750
- [Derived] Thumbigere-Math V, Alqadi A, Chalmers NI, Chavez MB, Chu EY, Collins MT, Ferreira CR, FitzGerald K, Gafni RI, Gahl WA, Hsu KS, Ramnitz MS, Somerman MJ, Ziegler SG, Foster BL. Hypercementosis Associated with ENPP1 Mutations and GACI. J Dent Res. 2018 Apr;97(4):432-441. doi: 10.1177/0022034517744773. Epub 2017 Dec 15. PMID 29244957
- [Derived] Gunay-Aygun M, Zivony-Elboum Y, Gumruk F, Geiger D, Cetin M, Khayat M, Kleta R, Kfir N, Anikster Y, Chezar J, Arcos-Burgos M, Shalata A, Stanescu H, Manaster J, Arat M, Edwards H, Freiberg AS, Hart PS, Riney LC, Patzel K, Tanpaiboon P, Markello T, Huizing M, Maric I, Horne M, Kehrel BE, Jurk K, Hansen NF, Cherukuri PF, Jones M, Cruz P, Mullikin JC, Nurden A, White JG, Gahl WA, Falik-Zaccai T. Gray platelet syndrome: natural history of a large patient cohort and locus assignment to chromosome 3p. Blood. 2010 Dec 2;116(23):4990-5001. doi: 10.1182/blood-2010-05-286534. Epub 2010 Aug 13. PMID 20709904
- [Derived] Maynard DM, Heijnen HF, Gahl WA, Gunay-Aygun M. The alpha-granule proteome: novel proteins in normal and ghost granules in gray platelet syndrome. J Thromb Haemost. 2010 Aug;8(8):1786-96. doi: 10.1111/j.1538-7836.2010.03932.x. Epub 2010 May 27. PMID 20524979
- [Derived] Huizing M, Dorward H, Ly L, Klootwijk E, Kleta R, Skovby F, Pei W, Feldman B, Gahl WA, Anikster Y. OPA3, mutated in 3-methylglutaconic aciduria type III, encodes two transcripts targeted primarily to mitochondria. Mol Genet Metab. 2010 Jun;100(2):149-54. doi: 10.1016/j.ymgme.2010.03.005. Epub 2010 Mar 16. PMID 20350831
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1976-HG-0238.html